CLINICAL TRIAL: NCT03053206
Title: RESPONSE TO CYTARABINE, DAUNORUBICIN AND ETOPOSIDE (ADE) AT FIRST RELASPE IN CHILDHOOD AML
Brief Title: A Prospective, Interventional Study Assessing Response to Cytarabine, Daunorubicin and Etoposide (ADE) for First Relapse of Paediatric Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, ARUN GARG, MD, DM, SENIOR RESIDENT, All India Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IECPG-660/22.12.2016
Record Dates: First submitted 2017-02-07; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Acute Myeloid Leukemia, in Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — DAV regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADE arm (Experimental): ADE arm
  Cytarabine (100mg/m2 d1-d10 BD), Daunorubicin (50mg/m2 d1-d3) and Etoposide (100 mg/m2 d1-5) over a period of 10 days
  Interventions: Drug: ADE Protocol

INTERVENTIONS:
Drug: ADE Protocol — ADE chemotherapy
  Cytarabine (100mg/m2 d1-d10 BD), Daunorubicin (50mg/m2 d1-d3) and Etoposide (100 mg/m2 d1-5) over a period of 10 days

SUMMARY:
One-third to one-half of patients with AML relapse and in general relapsed AML patients have a poor prognosis. The treatment of relapsed AML consists of induction chemotherapy followed by Allogenic Stem Cell Transplant (ASCT). However, at present there is no standard salvage chemotherapy regimen for relapsed AML, as no study has shown any one regimen to be significantly superior. Anthracyclines, Fludarabine, Etoposide and cytarabineare active agents in AMLand have been used as monotherapy and in combination in refractory and relapsed AML patients. According to previous studies the present CR rate of different regimens ranges from 50-70%. A retrospective analysis (unpublished) conducted at IRCH, AIIMS on relapsed AML patients treated with ADE (Cytarabine, Daunorubicin and Etoposide) chemotherapy showed the CR rates of approximately 70%. Therefore, we have planned this study to test the efficacy and toxicity of ADE induction chemotherapy in relapsed AML patients in a prospective manner.

ELIGIBILITY:
Inclusion Criteria:

1. Either gender with age ≤18 years at initial diagnosis
2. AML(non-M3) patients at first relapse (medullary)

Exclusion Criteria:

1. Primary refractory AML &secondary AML
2. More than or equal to 2 relapses of AML
3. Symptomatic cardiac dysfunction (CTCAE Grade 3 or 4)
4. Active infection(pneumonia etc.)
5. Any other organ dysfunction (CTCAE Grade 4)
6. Patients not willing to consent for the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-02-15 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
complete remission (CR) rate | Day 28 ± 7 of treatment or after recovery of blood counts whichever is earlier
  To assess the complete remission (CR) rate with the use of ADE chemotherapy in relapsed acute myeloid leukemia (AML) after first CR

SECONDARY OUTCOMES:
Event free survival (EFS) and overall survival(OS) | 2 year
  To determineevent free survival(EFS) and overall survival(OS)
toxicity of chemotherapy | Day 28 ± 7 of treatment
  To assess the toxicity of chemotherapy using CTCAE 4.0
clonal evolution | Day 28 ± 7 of treatment
  To evaluate clonal evolution using cytogenetics &RT-PCR panel
minimal residual disease (MRD) | Day 28 ± 7 of treatment or after recovery of blood counts whichever is earlier
  To assess minimal residual disease (MRD) by using flow cytometry
cardiac function | Day 28 ± 7 of treatment
  To evaluate cardiac function using 2 Dimensional Echocardiography

IPD SHARING:
Plan to Share IPD: No